CLINICAL TRIAL: NCT07105228
Title: Incidence of Retinal Vasculitis Among Patients Receiving Aflibercept: A US Real-World Evidence Study
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VGFTe-OD-2458
Record Dates: First submitted 2025-07-08; First posted 2025-08-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Retinal Vasculitis
Keywords: Anti-Vascular Endothelial Growth Factor (VEGF); Aflibercept; neovascular Age-related Macular Degeneration (nAMD); Diabetic Macular Edema (DME); Diabetic Retinopathy (DR); Macular Edema Following Retinal Vein Occlusion (RVO)
MeSH Terms: conditions — Retinal Vasculitis; Diabetic Retinopathy | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Patients: Patients ≥ 18 years of age, who received aflibercept 2mg IVT during the study period
  Interventions: Drug: aflibercept 2mg

INTERVENTIONS:
Drug: aflibercept 2mg — No study-specific interventions administered in this observational study
  Other Names: Eylea®

SUMMARY:
This study will describe and estimate the incidence of Retinal Vasculitis (RV) events among patients and patient eyes receiving aflibercept intravitreal (IVT) (Eylea®, aflibercept 2mg) therapy in US clinical practice.

The main objective is to describe demographic and clinical characteristics of patients receiving aflibercept 2mg injections, to estimate the incidence of RV and RV plus Intraocular Inflammation (IOI) following aflibercept 2mg injections and to describe characteristics of RV cases.

DETAILED DESCRIPTION:
This study is purely descriptive using US claims data from Komodo Healthcare Map.

ELIGIBILITY:
Inclusion Criteria for Patient Population:

1. All aflibercept injections identified by the Healthcare Common Procedure Coding System (HCPCS) or National Drug Code (NDC) from January 1, 2017, to February 29, 2024, as recorded in the Komodo close claims database.

Key Exclusion Criteria:

1. Aflibercept injections with unspecified laterality will be excluded
2. Aflibercept injections from individuals aged <18 years or those with unknown age on the injection date will be excluded
3. Patient-eyes with a diagnosis of RV in the same eye as the aflibercept injection or with unspecified laterality within 12 months (365 days) prior to index date (inclusive), as defined in the protocol
4. Patient-eyes that do not meet the continuous enrollment requirement will be excluded
5. Aflibercept injections will be excluded if there is ≥1 other anti-VEGF injection administered on the same date

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will represent patients and patient-eyes who initiate aflibercept 2 mg injections
Sampling Method: Non-Probability Sample
Enrollment: 290000 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of RV events | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 7 years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-10) diagnosis codes
Incidence of RV plus IOI events | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 7 years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-10) diagnosis codes
Demographics characteristics | 12 months prior to the index date
  Demographics include: sex, age, race/ethnicity, insurance, geographic area
Clinical characteristics: Number of participants with different retinal disease diagnosis categories | 12 months prior to the index date
  Retinal disease categories: nAMD, DME, DR w/o DME, or macular edema following retinal vein occlusion [MEfRVO])
Clinical characteristics: Mean Charlson Comorbidity Index (CCI) score | 12 months prior to the index date
  The Charlson Comorbidity Index (CCI) is a method used to categorize comorbidities based on International Classification of Diseases (ICD) diagnosis codes. A score of 0 indicates that no comorbidities were found, while higher scores correspond to increased predicted mortality
Clinical characteristics: Summary of comorbidities reported as number of participants with different categories | 12 months prior to the index date
  Different comorbidity categories: Syphilis, Herpesviridae, Toxoplasmosis, Tuberculosis, Systemic lupus erythematosus, Multiple sclerosis, Behçet's disease, Cardiovascular disease, Hypertension, Diabetes, Hypercholesterolemia
Clinical characteristics: Number of participants with prior anti-VEGF treatment | 12 months prior to the index date

SECONDARY OUTCOMES:
Incidence of RV plus RO | During the 60-Day at-risk period following aflibercept 2 mg IVT, up to approximately 7 years
  Incidence will be defined as the number of events during the at-risk period divided by the total number of injections, identified using international classification of diseases (ICD-10) diagnosis codes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, Tarrytown, New York, United States